CLINICAL TRIAL: NCT04727541
Title: Neoadjuvant Bintrafusp Alfa in Patients With Resectable Biliary Tract Cancer
Acronym: NEOBIL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on results of another phase II study with bintrafusp alfa in combination with gemcitabine plus cisplatin, that was discontinued as it was unlikely to meet the primary endpoint of OS, the recruitment for this study was stopped prematurely.
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Merck Serono GmbH, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-HEP-0120; 2020-002605-25 (EudraCT Number); MS200647_0075 (Other Grant/Funding Number: Merck Healthcare KGaA)
Record Dates: First submitted 2021-01-25; First posted 2021-01-27 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy with Bintrafusp alfa (Experimental): 1200 mg of Bintrafusp alfa will be administered by intravenous infusion every 2 weeks for a total of 2 dosages (Q2W). Subsequently, the surgery will be performed.
  Interventions: Drug: Bintrafusp alfa

INTERVENTIONS:
Drug: Bintrafusp alfa — Neoadjuvant therapy with bintrafusp alfa
  Other Names: MSB0011359C, M7824

SUMMARY:
The NEOBIL study aims to investigate the feasibility, safety and efficacy of neoadjuvant Bintrafusp alfa in patients with resectable biliary tract cancer.

DETAILED DESCRIPTION:
The only curative therapy for biliary tract cancer (BTC) is resection. However, recurrence rates are very high with a median recurrence-free survival (RFS) time of 18 months with adjuvant chemotherapy. Bintrafusp alfa is a bifunctional fusion protein targeting TGF-β and PD-L1 that has shown promising activity in a second-line phase I BTC study. The neoadjuvant treatment approach is not a current standard in biliary tract cancer, but it is an accepted and frequently applied treatment strategy in other resectable and borderline-resectable cancers such as lung, gastric and rectal cancer. The hypothesis is that Bintrafusp alfa leads to a major pathological response in 30% of resectable BTC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent granted prior to initiation of any study-specific screening procedures
2. Biliary tract cancer, confirmed by histopathology, cytopathology is not sufficient
3. Resectable disease limited to the liver assessed by an interdisciplinary tumor board involving a hepatobiliary surgeon; no prior systemic therapy
4. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
5. Age ≥ 18 years
6. Performance status ECOG 0-1
7. Normal organ and bone marrow function defined as:

   * Hematopoetic: absolute neutrophil count ≥1,500/mm3, platelet count ≥ 100,000/mm3,
   * Hemoglobin ≥9 g/dL
   * Normal international normalized ratio (INR), PT ≤ 1.5 x ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
   * Hepatic: AST ≤5 x ULN, ALT ≤ 5 x ULN, and bilirubin ≤ 3.0 x ULN.
   * Renal: Creatinine level ≤1.5 x ULN or estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
8. Special medical conditions and comorbidities:

   * Maximum Child Pugh stage A in patients with cirrhosis
   * HIV: stable on ART for at least 4 weeks, no documented evidence of multi-drug resistance, viral load of < 400 copies/mL and CD4+ T-cells ≥ 350 cells/µL.
   * HBV infection: participant on a stable dose of antiviral therapy, HBV viral load below the limit of quantification.
9. Women of childbearing potential must have a negative serum or highly sensitive urine pregnancy test performed within 7 days prior to the first dose of IMP.
10. Women of childbearing potential (WOCBP) must use HIGHLY EFFECTIVE method(s) of contraception to avoid pregnancy for the duration of study treatment and further 2 months after the last dose of IMP.
11. Male participants who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception or to abstain from sexual activity and will be instructed to adhere to either method from the time of first dose until 125 days after the last dose of investigational product. In addition, male subjects must be willing to refrain from sperm donation during this time. Azoospermic men do not require contraception.

Exclusion Criteria:

1. Metastatic disease
2. Prior surgery, systemic therapy, radiation therapy, chemoradiation, transarterial chemoembolisation (TACE), Radiofrequency ablation (RFA) or selective intraarterial Radiotherapy (SIRT) for treatment of CCA. NOTE: Laparoscopy for diagnostic procedures is allowed.
3. Drug or alcohol addiction, medical or psychological condition that may interfere with the patient´s participation in the study
4. Participation in another clinical trial with any investigational study drug (whatever the use, curative, prophylactic or diagnostic intent) within 30 days prior to enrollment
5. Pregnancy or breast feeding women
6. Regulatory and ethical criteria:

   * Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities [§ 40 Abs. 1 S. 3 Nr. 4 AMG].
   * Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].
7. IMMUNOSUPRESSANTS: "Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)."
8. AUTOIMMUNE DISEASE: "Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible."
9. PREVIOUS MALIGNANT DISEASE: within the last 3 years except for a. superficial/non-invasive bladder cancer, or basal or squamous cell carcinoma in situ treated with curative intent; b. endoscopically resected GI cancers limited to the mucosal layer without recurrence in > 1 year.
10. INFECTIONS: "Active infection requiring systemic therapy. "
11. VACCINATION: has received or will receive a live vaccine within 30 days prior to the first administration of study intervention. Seasonal flu vaccines that do not contain a live virus are permitted. Locally approved COVID vaccines are permitted.
12. HYPERSENSITIIVTY TO BINTRAFUSP ALFA: "Known severe hypersensitivity [Grade ≥ 3 NCI CTCAE 5.0]) to investigational product bintrafusp alfa or any component in its formulations, any history of anaphylaxis, or recent, within 5 months, history of uncontrollable asthma.
13. CARDIOVASCULAR DISEASE: "Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication."
14. BLEEDING: "history of bleeding diathesis or recent major bleeding events (i.e. Grade ≥ 2 bleeding events in the month prior treatment)
15. Other severe acute or chronic medical conditions: "including drug-induced interstitial lung disease (ILD) or participant has had a history of drug-induced pneumonitis that has required oral or IV steroids", and/or other diseases, which in the opinion of the Investigator might impair the participant's tolerance for the study or ability to consistently participate in study procedures.
16. Uncontrolled diabetes as defined by HbA1c > 10.0 %.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Major Pathologic Response (MPR) measured in the surgically resected tumor | 24 months
  Response to neoadjuvant treatment will be determined according to the Becker score. MPR is defined by a Becker grade of 1 (1a or 1b), namely at least < 10% of viable tumor.

SECONDARY OUTCOMES:
Tumor Response | 24 months
  Tumor Response according to RECIST1.1
Rate of Resectability | 24 months
  Rate of Resectability in biliary tract cancer patients
Adverse events according to CTCAE V5 | 24 months
Adverse Events of Special Interest | 24 months
  Postoperative wound infections, impaired wound healing, wound dehiscence, prolongation of post-op hospitalization beyond 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Waidmann, Prof.Dr., Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (2):
- Germany (2):
  - Universitätsklinikum RWTH Aachen - Klinik für Allgemein-, Viszeral- und Transplantationschirurgie, Aachen
  - Universitätsklinikum Frankfurt - Medizinische Klinik 1, Frankfurt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de/
- See also: Description AIO-Studien-gGmbH — http://www.aio-portal.de/